CLINICAL TRIAL: NCT02014662
Title: A Pilot Study to Measure Force Recovery and Protein Synthetic Rates After Unilateral Eccentric Exercise in Healthy Males Volunteers Unaccustomed to Eccentric Exercise
Brief Title: A Methodology Study to Assess Muscle Damage After Eccentric Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200794
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Tendon Injuries
Keywords: Muscle function, Muscle damage and recovery, Eccentric exercise, Muscle soreness, Protein synthesis
MeSH Terms: conditions — Tendon Injuries; Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Healthy subjects aged 18 to 35 years
  Interventions: Other: Eccentric exercise

INTERVENTIONS:
Other: Eccentric exercise — Each subject will perform eccentric exercise against a predefined personal maximal strength of their non-dominant leg on day 1. Changes on strength, biomarker concentrations and muscle protein synthesis during damage and recovery will be measured over 22 days.

SUMMARY:
An isolated bout of unaccustomed maximal eccentric exercise is associated with muscle force loss for 2-4 days, mild reversible muscle tenderness, and ultra-structural damage to the muscle fibers, elevation of muscle proteins in serum, and a detriment in range of motion. This single center, pilot study is designed to optimize conditions for the robust measurement of functional deficits after muscle damage and to identify markers of repair over 22 days to inform future intervention studies. The primary measure will be limb force (assessed electronically from the ergometer), previous studies have demonstrated that functional measures return fairly rapidly, usually between 2-4 days. Additionally, several biomarkers of muscle function will be measured over 22 days, as well as changes in protein synthesis in biopsy samples Deuterium-labelled water (D2O) will be consumed by all study participants from Day-3 through Day 22 to aid in quantifying newly synthesized proteins.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 35 years of age inclusive, at the time of signing the informed consent, not on a regular exercise program.
* Body Mass Index (BMI) 18-27 kilogram per meter square (kg/m^2) with waist circumference <96 centimeter (cm).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Based on single or averaged corrected QT interval (QTc) (Bazzett [QTcB] or Fredericia [QTcF]) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QTc <450 milliseconds (msec); or QTc < 480 msec in subjects with Bundle Branch Block.
* At least a 1year history of no regular (2-3 times per week) exercise and no heavy exertion within past week.

Exclusion Criteria:

* History of keloid scarring
* History of dizziness or vertigo
* History of bleeding disorders or elevated partial thromboplastin time/international normalized ratio (PTT/INR) at screening, or currently on anticoagulants
* Taking anti-inflammatory, glucocorticoid or other pain medication more than 2 times per week over the previous month.
* Taking regular statin medication.
* Herbal supplement use
* History of smoking or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of drug or alcohol abuse within 5 years prior to the Screening Period.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 gram (gm) of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to local anesthetics.
* History of sensitivity to any drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation

Criteria Based Upon Diagnostic Assessments:

* A positive pre-study drug/alcohol screen.

Other Criteria:

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2014-07-02 (Actual); Study Completion 2014-07-02 (Actual)

PRIMARY OUTCOMES:
Change and percent change in maximal leg isometric strength from the baseline up to three weeks after eccentric exercise | Day 1, 2, 3, 4, 6, 8, 11, 17 and Day 22
  Muscle strength is a measure the amount of force produced during a maximal voluntary contraction. Strength will be assessed by a maximal isometric (fixed length) contraction.

SECONDARY OUTCOMES:
Change in peak torque and total work performed over the course of 10 consecutive, maximal isokinetic knee extension and flexion contractions | Day 1, 2, 3, 4, 6, 8, 11, 17 and Day 22
  Each subject will be asked to produce 10 consecutive, maximal isokinetic knee extension and flexion contractions through the full range of motion with the exercised leg on an ergometer
Patient pain assessment using a visual analog scale | Day 1, 2, 3, 4, 6, 8, 11, 17 and Day 22
  Leg pain will be assessed for the exercised leg with a visual analog scale (0-100 mm) before and up to three weeks after eccentric exercise
Change in degree of motion | Day 1, 2, 3, 4, 6, 8, 11, 17 and Day 22
  Each subject will be asked to attempt to move the exercised leg through a full range of motion with zero resistance from baseline up to three weeks after eccentric exercise
Change in plasma CPK and aldolase | Day 1, 2, 3, 4, 6, 8, 11, 17 and Day 22
  Blood sample will be collected to assess CPK and aldolase from baseline and up to three weeks after eccentric exercise
Change in plasma markers | Day 1, 2, 3, 4, 6, 8, 11, 17 and Day 22
  Blood sample will be collected to assess blood inflammatory markers including, but are not limited to, tissue necrosis factor alpha (TNFalpha), interleukin (IL) 1 beta, IL6, IL8, IL10, chemokine ligand (CCL)7, complement 3a (C3a), granulocyte macrophage colony stimulating factor (GM-CSF), and c-reactive protein (CRP) from baseline and up to three weeks after eccentric exercise

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

REFERENCES:
- See also: Results for study 200794 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200794?search=study&search_terms=200794#rs